CLINICAL TRIAL: NCT04155671
Title: A Phase 2 Study of POF(Paclitaxel/Oxaliplatin/5-Fluorouracil/Leucovorin) Versus FOLFOX Plus Intraperitoneal Paclitaxel as a First-line Treatment in Advanced Gastric Cancer With Peritoneal Metastases
Brief Title: POF Versus FOLFOX Plus IP Paclitaxel in AGC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF-018
Record Dates: First submitted 2019-10-31; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POF (Experimental): The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days. The combined chemotheraphy will be treated for 9 circle. then，the capetabine was allowed
  Interventions: Drug: POF
- FOLFOX plus PAC(ip) (Experimental): The regimen consisted of oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2) plus paclitaxel (80 mg/m2) intra-peritoneally.Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  Interventions: Drug: FOLFOX plus PAC(ip)

INTERVENTIONS:
Drug: POF — Paclitaxel plus Oxaliplatin plus Leucovorin plus 5-FU
  Arms: POF
Drug: FOLFOX plus PAC(ip) — FOLFOX plus intraperitoneally paclitaxel
  Arms: FOLFOX plus PAC(ip)

SUMMARY:
The aim of this study was to compare the efficacy and safety of intravenous or intraperitoneal paclitaxel plus FOLFOX as first-line treatment in AGC with peritoneal metastases, a phase II Clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* Patients must have histologically or cytologically confirmed metastatic or unresectable gastric or gastroesophageal junction (GEJ) adenocarcinoma. GEJ adenocarcinoma may be classified according to Siewert's classification type I, II, or III
* Histological documentation of local recurrence or metastasis is strongly encouraged, unless the risk of such a procedure outweighs the potential benefit of confirming the metastatic disease.
* If no histologic confirmation, then the metastases or recurrence will require documentation by a 2nd radiographic procedure (eg. PET/CT scan or MRI in addition to the CT scan). If the imaging procedure does not confirm recurrent or metastatic disease, biopsy confirmation will be required.
* Patients must have ascites or peritoneal carcinomatosis confirmed by image (CT or MR or US or others) operation.
* Patients may have received no prior chemotherapy for metastatic or unresectable disease. Patients may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if more than 6 months have elapsed between the end of adjuvant therapy and registration.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
* An expected survival of ≥ 3 months;
* Major organ function has to meet the following criteria; (1) For results of blood routine test:
* Hemoglobin (HB) ≥ 80g / L,
* ANC(absolute neutrophil count) ≥ 1.5 × 109 / L,
* PLT(blood platelet) ≥ 75 × 109 / L, (2) For results of biochemical tests:
* BLT（total bilirubin） ≤ 1.25 times the upper limit of normal (ULN),
* ALT(Alanine aminotransferase) and AST(aspartate aminotransferase ) ≤ 2.5 × ·ULN, liver metastases, if any, the ALT and AST≤ 5 × ULN,
* Serum Cr（creatinine）≤1ULN, Endogenous creatinine clearance rate >50ml/min;
* The patient has a PT（prothrombintime） (INR international normalized ratio) < or = to 1.5 and an PTT（Partial Thromboplastin Time）< than or = to 3 seconds above the upper limits of normal if the patientia t is not on anticoagulation. ·If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:
* The patient must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW(Low molecular weight) heparin
* The patient must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices)
* Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Ability to understand informed consent and signing of written informed consent document prior to initiation of protocol therapy.

Exclusion Criteria:

- Patients who have received previous chemotherapy for the treatment of metastatic or unresectable gastric or GEJ adenocarcinoma are ineligible.

* Patients who have received previous pre- or post-operative chemotherapy or chemoradiation are ineligible if therapy was completed less than 6 months prior to study registration. Patients must have recovered from adverse events from any previous therapy.
* Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
* Patients with brain or central nervous system metastases, including leptomeningeal disease.
* Pregnant (positive pregnancy test) or breast feeding.
* Serious, non-healing wound, ulcer, or bone fracture.
* Significant cardiac disease as defined as:

unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.

* History of a stroke or CVA within 6 months
* Clinically significant peripheral vascular disease.
* Inability to comply with study and/or follow-up procedures.
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | 12 months
  The length of time from enrollment until the time of death

SECONDARY OUTCOMES:
Adverse Event（AE） | 6month
  Adverse Event according to NCI CTCAE 5 criteria
Objective Overall Response Rate (ORR) | 6month
  Clinical response of treatment according to RESIST v1.1 criteria

IPD SHARING:
Plan to Share IPD: Undecided